CLINICAL TRIAL: NCT02591498
Title: Computerized Cognitive Training for Schizophrenia in Brazil
Acronym: CCTSB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Associate professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R03TW009002-01 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2015-10-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia
Keywords: cognitive training
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auditory (Active Comparator): Administration of 40 hours of auditory training exercises
  Interventions: Behavioral: Computerized cognitive training
- Visual (Active Comparator): Administration of 40 hours of visual training exercises
  Interventions: Behavioral: Computerized cognitive training
- Video Games (Placebo Comparator): Administration of 40 hours of commercial video games
  Interventions: Behavioral: Computerized cognitive training

INTERVENTIONS:
Behavioral: Computerized cognitive training

SUMMARY:
The purpose of this study is to investigate the effect of a neuroplasticity-based computerized cognitive training for people with schizophrenia in the Brazilian population.

DETAILED DESCRIPTION:
Cognitive impairments are important determinants of functional outcome in schizophrenia, which are inadequately treated by antipsychotic medication. Neuroplasticity based computerized cognitive trainings have been emerging for the last two decades and are an attempt to help patients with their cognitive impairments and global functioning.

The aim of this study is to perform a computerized cognitive training to improve attention, concentration, learning, clinical symptoms and quality of life in patients. The investigators are interested in testing the differential efficacy between a specific visual versus auditory computerized cognitive training and explore the biological markers that may be involved in these neuroplasticity based training processes.

The investigators will conduct a 40 hours computerized, adaptable, perception specific, cognitive training program in patients with schizophrenia. Patients will come for 1 hour, daily, and perform a visual or auditory training, or control games for about 2 months. Visual and auditory exercises are chosen to be the equivalent of one another and target cognitive domains such as divided attention, working memory and social cognition. Clinical, cognitive, emotional and biomarker data will be collected before the training, half way through, and after the training, to assess progress in several aspects of their functioning and biology.

The investigators hypothesize visual and auditory trainings will be effective as compared to the control games. They also expect that auditory training to be more efficient compared to the visual training because it targets sensory functions that are mostly impaired in schizophrenia, due to auditory hallucinations patients experience. The investigators also hypothesize that both trainings will improve clinical symptoms and quality of life. On a more exploratory analysis, the investigators expect to identify new biological markers of cognitive neuroplasticity, which they expect will differentiate visual and auditory paths.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia or schizoaffective disorder based on DSM-IV criteria
* age 18- 60 years
* Portuguese as primary language (learned before age 12)
* no major medical or neurological disorder that precludes participation in the study

Exclusion Criteria:

* IQ score <70
* active substance dependence (DSM-IV criteria)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Global cognition score change | through study completion, an average of 1 year
  The global cognition score is a composite measure from the MATRICS (Measurement And Treatment Research to Improve Cognition in Schizophrenia) Consensus Cognitive Battery tests

SECONDARY OUTCOMES:
Processing speed score change | through study completion, an average of 1 year
  Processing speed score will be measured using the Motor task from CANTAB (Cambridge Neuropsychological Test Automated Battery) test and the category fluency
Attention score change | through study completion, an average of 1 year
  Attention score will be measured using the Reaction time test and Rapid visual processing CANTAB tests
Working memory score change | through study completion, an average of 1 year
  Working memory will be measured using the Spatial working memory CANTAB test and the digit backward
Verbal memory and learning score change | through study completion, an average of 1 year
  Verbal memory and learning score will be measured using the Hopkins verbal learning test
Visuospatial memory and learning score change | through study completion, an average of 1 year
  Visuospatial memory and learning score will be measured using the brief visuospatial memory test
Reasoning and problem solving score change | through study completion, an average of 1 year
  Reasoning and problem solving score will be measured using the Stockings of Cambridge CANTAB test
Reward task score change | through study completion, an average of 1 year
  Reward task score will be measured using the reward task (adapted from Graham Murray)
Emotional inhibition control score change | through study completion, an average of 1 year
  Emotional inhibition control score will be measured using the Affective go no go CANTAB test
Biological markers from the glutamatergic system change | through study completion, an average of 1 year
  Biological markers from the glutamatergic system will be measured using High profile liquid chromatography
Genes of neuroplasticity | through study completion, an average of 1 year
  Genes of neuroplasticity will be measured using candidate genotyping and Genome wide analysis
Eotaxin 1 change | through study completion, an average of 1 year
  Levels of eotaxin 1 will be measured using ELISA kit
Prepulse inhibition change | through study completion, an average of 1 year
  Prepulse inhibition will be measured via eye muscle reaction to sound
Eye-tracking change | through study completion, an average of 1 year
  Eye-tracking will be measured via an infrared camera while patients do cognitive tests
Electroencephalogram (EEG) change | through study completion, an average of 1 year
  EEG will be measured with electrodes on the surface of the skull while patients do cognitive tests
motivation scores change | through study completion, an average of 1 year
  Motivation scores will be measured with an interview and the Behavior Inhibition/Activation Scale questionnaire
Depression score change | through study completion, an average of 1 year
  Depression score will be measured using the Hamilton - Depression questionnaire
Anxiety score change | through study completion, an average of 1 year
  Depression score will be measured using the Hamilton - Anxiety questionnaire
Mood scores change | through study completion, an average of 1 year
  mood scores will be measured using the Visual analogue scale (Norris 1971)
Positive and negative syndrome scale score change | through study completion, an average of 1 year
  Clinical score will be measured using the Positive and Negative Syndrome Scale for Schizophrenia
Quality of Life change | through study completion, an average of 1 year
  Quality of life will be measured using the World Health Organization of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Panizzutti, M.D., Ph.D., Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil